CLINICAL TRIAL: NCT06790979
Title: Wearable Device-Based Analysis of the Relationship Between Sleep Patterns and Clinical Prognosis in Patients With Mild to Moderate Traumatic Brain Injury
Brief Title: Wearable Device-Based Analysis of the Relationship Between Sleep Patterns and Clinical Prognosis in Patients With Traumatic Brain Injury
Status: Recruiting | Type: Observational
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Jingchao Zhou
Record Dates: First submitted 2025-01-18; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-11

CONDITIONS: Traumatic Brain Injury (TBI); Concussion, Initial Encounter
Keywords: Traumatic brain injury; Sleep; Prognosis of trauma; Wearable devices
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In patients with traumatic brain injury, post-traumatic sleep patterns have the potential to impact clinical prognosis. While some progress has been made in the study of sleep and prognosis in patients with traumatic brain injury, there is still lack of research on the relationship between sleep and clinical prognosis in post-traumatic patients due to differences in study design, patient age, severity of trauma, and definitions of sleep disorders. Additionally, the primary data collection methods employed in most studies have been self-reported sleep assessments, which are subject to potential biases and inaccuracies. Therefore, explore the impact of sleep patterns on clinical prognosis in post-traumatic patients, with potential to advance our comprehension of recovery outcomes in this patient group.

ELIGIBILITY:
Inclusion Criteria:

1. 18~60 years old.
2. The patient had no sleep disturbance problems prior to traumatic brain injury.
3. The patient has a definite diagnosis of traumatic brain injury and the Glasgow score is >8.
4. The patient had abnormal imaging scans.
5. It has complete preclinical data.

Exclusion Criteria:

1. Patients with a previous history of traumatic brain injury, mental illness, alcohol abuse or sleep disorders.
2. Patients admitted for surgical intervention.
3. Patients with a combination of other heavy visceral injuries.
4. Women during pregnancy and lactation.
5. The patents' use of medications that interfere with sleep

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Qualified inpatients hospitalized in our hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Change of cognitive function | 1st day and 30th day
  The use of MOCA to measure cognitive function in patients with TBI.
Change of executive function | 1st day and 30th day
  The use of the TMT-B to measure executive function in patients with TBI.

CONTACTS AND LOCATIONS:
Overall Officials: Zhanfeng Niu, Doctor, Study Director — General Hospital of Ningxia Medical University
Locations (1):
- The General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China